CLINICAL TRIAL: NCT03017157
Title: Subclinical Hypothyroidism and Acute Anterior Myocardial Infarction: Is it Cardio-protective or Not?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0096-16-HYMC
Record Dates: First submitted 2016-12-21; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Heart Injuries
MeSH Terms: conditions — Heart Injuries | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Anterior Myocardial Infarction: Patients who have suffered anterior myocardial infarction in our hospital
  Interventions: Other: Echo-cardiogram; Other: Blood test

INTERVENTIONS:
Other: Echo-cardiogram — Patients will undergo echo-cardiogram to determine improvement in their heart function and this will be compared to thyroid function
Other: Blood test — Blood test to determine thyroid function

SUMMARY:
The study plans to investigate whether recovery of the heart function after acute anterior myocardial infarction is dependent upon improvement in thyroid gland functioning.

ELIGIBILITY:
Inclusion Criteria:

* Have suffered anterior myocardial infarction

Exclusion Criteria:

* Do not receive thyroid treatment
* No history of ischemic heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered anterior myocardial infarction who have been hospitalized in our hospital's cardiac unit.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Ejection Fraction Improvement | 40 days
  Improvement in ejection fraction as shown in echo-cardiogram
Improvement in thyroid function | 40 days
  Thyroid stimulating hormone (TSH) level will be normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No